CLINICAL TRIAL: NCT03021382
Title: Comparisons of Morphological Measurement Between Coronary Computed Tomography and Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Kobe University (Industry)
Collaborators: HeartFlow, Inc. (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, Department of Internal Medicine, Kobe University Graduate School of Medicine, Kobe University
Other Study IDs: No.160040
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- severity of calcification: All vessels were divided into tertile groups according to the severity of coronary calcification evaluated by the Agatston score.
  Interventions: Other: data collection, non-intervention
- minimal lumen diameter (MLD) ≥1.0 mm: All lesions were divided according to an MLD ≥1.0 mm, and <1.0 mm by OCT in order to isolate the lesions which an MLD below the OCT catheter size.
  Interventions: Other: data collection, non-intervention

INTERVENTIONS:
Other: data collection, non-intervention

SUMMARY:
The objective of this study is to evaluate the precision of semi-automated lumen boundary identification from coronary computed tomography angiography (cCTA) by current version of HeartFlow software and the impact on fractional flow reserve (FFRCT) by using optical coherence tomography (OCT) as reference standard.

DETAILED DESCRIPTION:
Analysis of cCTA and OCT was conducted under blind in independent organizations.

After unblinding the cCTA and OCT case identification number, the OCT image was co-registered to cCTA data.

After co-registration of cCTA and OCT lesion locations, the minimal lumen area (MLA) was detected with both modalities. FFROCT was calculated using OCT-updated models in which cCTA-based lumen geometry was replaced by OCT-based lumen geometry.

Lesions were grouped according to their severity of calcification (using Agatston score) and minimum lumen diameter.

ELIGIBILITY:
Inclusion Criteria:

- Patients who underwent cCTA prior to coronary angiography and OCT within 6 months.

Exclusion Criteria:

1. Prior coronary artery bypass graft (CABG) surgery
2. Contraindication to beta blocker agents or nitrates
3. Tachycardia or significant arrhythmia
4. Impaired chronic renal function (eGFR <30)
5. Subjects with known anaphylactic allergy to iodinated contrast material
6. Pregnancy or unknown pregnancy status in subject of childbearing potential
7. Cases with poor OCT or CCTA image for analyzing

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 72 vessels in 57 patients
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Correlation between cCTA and OCT for MLA measurements | Immediately after OCT scan

SECONDARY OUTCOMES:
Correlation between FFRCT and FFROCT | Immediately after OCT scan
Impact of calcification on the agreement of MLA between OCT and cCTA measurement | Immediately after OCT scan
Impact of calcification on the agreement of FFR between OCT and cCTA | Immediately after OCT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Kobe University Graduate School of Medicine, Department of Cardiology, Kobe, Hyōgo, Japan